CLINICAL TRIAL: NCT05119920
Title: Multicenter, Randomized, Double-Masked, Placebo-Controlled, Parallel Group Phase 2 Trial Evaluating the Safety and Efficacy of Pilocarpine Ophthalmic Topical Cream BID for the Treatment of Signs and Symptoms of Dry Eye Disease
Brief Title: Safety and Efficacy of Pilocarpine Ophthalmic Topical Cream for the Treatment of Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ILUT-401-DED
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Dry Eye Disease; Kerato Conjunctivitis Sicca
Keywords: Dry eye syndromes; Eye diseases; Corneal diseases; Keratoconjunctivitis; Pilocarpine
MeSH Terms: conditions — Dry Eye Syndromes; Eye Diseases; Corneal Diseases; Keratoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pilocarpine Ophthalmic Topical Cream, Dose 1 (Experimental): Pilocarpine Ophthalmic Topical Cream, Dose 1
  Interventions: Drug: Pilocarpine Ophthalmic Topical Cream, Dose 1
- Pilocarpine Ophthalmic Topical Cream, Dose 2 (Experimental): Pilocarpine Ophthalmic Topical Cream, Dose 2
  Interventions: Drug: Pilocarpine Ophthalmic Topical Cream, Dose 2
- Pilocarpine Ophthalmic Topical Cream, Dose 3 (Experimental): Pilocarpine Ophthalmic Topical Cream, Dose 3
  Interventions: Drug: Pilocarpine Ophthalmic Topical Cream, Dose 3
- Placebo Ophthalmic Topical Cream (Placebo Comparator): Placebo Ophthalmic Topical Cream
  Interventions: Drug: Placebo Ophthalmic Topical Cream

INTERVENTIONS:
Drug: Pilocarpine Ophthalmic Topical Cream, Dose 1 — Pilocarpine Ophthalmic Topical Cream, Dose 1
  Other Names: GLK-301
  Arms: Pilocarpine Ophthalmic Topical Cream, Dose 1
Drug: Pilocarpine Ophthalmic Topical Cream, Dose 2 — Pilocarpine Ophthalmic Topical Cream, Dose 2
  Other Names: GLK-301
  Arms: Pilocarpine Ophthalmic Topical Cream, Dose 2
Drug: Pilocarpine Ophthalmic Topical Cream, Dose 3 — Pilocarpine Ophthalmic Topical Cream, Dose 3
  Other Names: GLK-301
  Arms: Pilocarpine Ophthalmic Topical Cream, Dose 3
Drug: Placebo Ophthalmic Topical Cream — Placebo Ophthalmic Topical Cream
  Other Names: Placebo
  Arms: Placebo Ophthalmic Topical Cream

SUMMARY:
This is a Multicenter, Randomized, Double-Masked, Placebo-Controlled, Parallel Group Phase 2 Trial Evaluating the Safety and Efficacy of Pilocarpine Ophthalmic Topical Cream for the Treatment of Signs and Symptoms of Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older at the Screening Visit
* Willing and able to provide written informed consent on the IRB/IEC-approved informed consent form
* Diagnosis of dry eye

Exclusion Criteria:

* Sensitivity or known allergy to pilocarpine or any of the other excipients of the formulation
* History of eczema, dermatitis or skin sensitivity to over-the-counter personal care products such as lotions, creams, makeup, soaps, etc.
* History of, or active iritis or uveitis in either eye
* Pre-existing retinal disease in either eye that may predispose subjects to retinal detachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in the VAS score at Day 28 visit. | Baseline and Day 28
  Mean change from baseline in the VAS score at Day 28 visit.
  Visual Analogue Scale from 0 (no discomfort) to 100 (maximal discomfort)
Mean change from baseline in Fluorescein Staining at the Day 28 visit. | Baseline and Day 28
  Mean change from baseline in Fluorescein Staining at the Day 28 visit.

SECONDARY OUTCOMES:
Mean change from baseline in the VAS score at the Day 4, 8, and 14 visits | Baseline and Days 4, 8, and 14
  Mean change from baseline in the VAS score at the Day 4, 8, and 14 visits
  Visual Analogue Scale from 0 (no discomfort) to 100 (maximal discomfort)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Glaukos Investigator, Chandler, Arizona
  - Glaukos Investigator, Sun City, Arizona
  - Glaukos Investigator, Glendale, California
  - Glaukos Investigator, Mission Hills, California
  - Glaukos Investigator, Newport Beach, California
  - Glaukos Investigator, Petaluma, California
  - Glaukos Investigator, Rancho Cordova, California
  - Glaukos Investigator, Grand Junction, Colorado
  - Glaukos Investigator, Fort Myers, Florida
  - Glaukos Investigator, Roswell, Georgia
  - Glaukos Investigator, St Louis, Missouri
  - Glaukos Investigator, Henderson, Nevada
  - Glaukos Investigator, Rochester, New York
  - Glaukos Investigator, Cranberry Township, Pennsylvania
  - Glaukos Investigator, Memphis, Tennessee
  - Glaukos Investigator, Nashville, Tennessee
  - Glaukos Investigator, Houston, Texas
  - Glaukos Investigator, San Antonio, Texas
  - Glaukos Investigator, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No